CLINICAL TRIAL: NCT04579536
Title: Effectiveness of Using a Light Curable Resin Modified Glass Ionmer Cement Varnish (Vanish XT) in Prevention of Occlusal Caries: a Randomized Controlled Clinical Trial
Brief Title: Effectiveness of Using (Vanish XT) in Prevention of Occlusal Caries: a RCT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: King Abdulaziz University (Other)
Responsible Party: Principal Investigator, Alaa M. Baik, paediatric dentist specialist, King Abdulaziz University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: Alaa Baik
Record Dates: First submitted 2020-10-06; First posted 2020-10-08 (Actual); Last update posted 2020-10-08 (Actual); Status verified 2020-10

CONDITIONS: Caries Prevention
Keywords: occlusal caries; Vanish XT varnish; Clinpro XT varnish; Light curable resin modified glass ionomer varnish; deep pits and fissures; newly erupted permanent first molars

STUDY DESIGN:
Intervention Model Description: The design of the study is a split-mouth, randomized controlled clinical trial in which the teeth are randomly assigned to be either in the test group or the control group in a 1:1 ratio. The control group: will be treated with 5% sodium fluoride (NaF) white varnish, oral hygiene instruction, and dietary counseling. The test group: will be treated with light curable resin modified glass ionomer (RMGI) varnish.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Triple blinding. Because of the nature of the material, the investigator who will apply the material to the occlusal surfaces will not be blinded to the group allocation. However, the investigators who will perform the clinical visual examination and the radiographic examination will be blinded to which group the teeth they are evaluating belongs. In addition, the statistician will be blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Study group (Experimental): This is the study group; it will consist of 84 first permanent molars. These molars will be sealed using light curing resin-modified glass ionomer varnish (ClinproTM XT Vanish, 3M ESPE, Dental Products, St. Paul, MN, USA). reapplication will be done after 3,6, 12, and 18 months.
  Interventions: Other: Light curable resin modified glass ionomer varnish
- Control group (Other): This group will consist of 84 first permanent molars. These molars will receive 5% Sodium Fluoride (NaF) with Tri-Calcium Phosphate topical varnish (Vanish White Varnish, 3M ESPE, Dental Products, St. Paul, MN, USA). These molars will serve as a control group. reapplication will be done after 3,6, 12, and 18 months.
  Interventions: Other: Vanish White Varnish

INTERVENTIONS:
Other: Light curable resin modified glass ionomer varnish — Light curing resin-modified glass ionomer varnish (ClinproTM XT Vanish, 3M ESPE, Dental Products, St. Paul, MN, USA) will be used to seal 84 first permanent molars at baseline, 3, 6, 12 and 18 months.
  Other Names: Vanish™ XT Extended Contact Varnish
  Arms: Study group
Other: Vanish White Varnish — 5% Sodium Fluoride (NaF) with Tri-Calcium Phosphate topical varnish (Vanish White Varnish, 3M ESPE, Dental Products, St. Paul, MN, USA) will be used on 84 first permanent molars at baseline, 3, 6, 12 and 18 months.
  Arms: Control group

SUMMARY:
Despite the continuous effort to prevent and treat dental caries, it continues to be one of the most common chronic diseases in both children and adults. Prevention and minimally intervention treatment by early detection of the lesion are becoming the new philosophy in managing dental caries. The prevalence of pit and fissure caries was found to be 90% of all dental caries in permanent molars. Moreover, the risk of caries development is higher soon after the tooth had erupted.

The purpose of the current study is; to evaluate the effectiveness of a resin-modified glass ionmer cement (Vanish XT) varnish in the prevention of occlusal caries and compare it to a fluoride varnish in newly erupted first permanent molars.

DETAILED DESCRIPTION:
material and method: The sample will comprise of 84 bilateral pairs of newly erupted first permanent molars in children with age of 6-9 years.This sample will be randomly selected after patient's screening from pediatric dentistry clinics at King Abdul-Aziz University Dental Hospital, Jeddah, Saudi Arabia. Informed written consent will be obtained from the parents prior to sampling.

Healthy children with all four first permanent molar will be included in the study. Children must have at least one pair of contralateral newly erupted first permanent molars free from caries. Teeth with deep pits and fissures free of caries, restorations, sealants, fracture, hypoplasia, or cracks will be included in the study.

The children who met the inclusion criteria will be enrolled in the trial after a signed consent form is obtained. Pairs of maxillary or mandibular first molars will be included so that one side will be randomly assigned to study group and the contralateral side to control group.

Study group: This group will consist of 84 first permanent molars. These molars will be sealed using light curing resin-modified glass ionomer varnish (ClinproTM XT Vanish, 3M ESPE, Dental Products, St. Paul, MN, USA)

Control group: This group will consist of 84 first permanent molars. These molars will receive 5% Sodium Fluoride (NaF) with Tri-Calcium Phosphate topical varnish (Vanish White Varnish, 3M ESPE, Dental Products, St. Paul, MN, USA). These molars will serve as a control group.

The clinical examination will be assessing the caries lesions at baseline and 3,6, 12, and 18 months by the trained and calibrated dentists' according to ICDAS II criteria (International Caries Detection and Assessment System). Teeth with deep pits and fissures, which scored 0 will be included in this study.

In addition, once the clinical examination is done, bitewing radiographs will be taken for each child on the first visit to diagnose caries at the baseline.

A child structured questionnaire to be completed by interviewing the parents (adopted from WHO Oral Health Questionnaire for Children) concerning the dental history of the child and oral hygiene habits will be given at the baseline and at each recall visit.

ELIGIBILITY:
Inclusion Criteria:

* Healthy children having no history of any systemic condition.
* Children must have all four first permanent molar.
* Children must have at least one pair of contralateral newly erupted first permanent molars free from caries.
* Teeth with deep pits and fissures (at high risk for caries).
* These molars should be free of caries, restorations, sealants, fracture, hypoplasia, or cracks.
* High caries risk children.

Exclusion Criteria:

* Children whom their parents refused to sign the consent form.
* Children older than 9 years old.
* Medically compromised children.
* Children having discolored grooves, restored, caries, or hypoplastic first permanent molars.
* Children having proximal caries in first permanent molars.
* Children whose antagonist teeth were extracted or not erupted.
* Children with a known acrylate allergy.
* Uncooperative children.

Ages: 6 Years to 9 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 84 (Estimated)
Dates: Start 2019-02-01 (Actual); Primary Completion 2020-02-01 (Actual); Study Completion 2021-07 (Estimated)

PRIMARY OUTCOMES:
caries development | 3 months
  To evaluate development of occlusal caries in newly erupted permanent first molars using the ICDAS after treating the surface with light curable RMGI varnish and compare it with contra-lateral teeth which received white varnish.
caries development | 6 months
  To evaluate development of occlusal caries in newly erupted permanent first molars using the ICDAS after treating the surface with light curable RMGI varnish and compare it with contra-lateral teeth which received white varnish.
caries development | 12 months
  To evaluate development of occlusal caries in newly erupted permanent first molars using the ICDAS after treating the surface with light curable RMGI varnish and compare it with contra-lateral teeth which received white varnish.
caries development | 18 months
  To evaluate development of occlusal caries in newly erupted permanent first molars using the ICDAS after treating the surface with light curable RMGI varnish and compare it with contra-lateral teeth which received white varnish.

CONTACTS AND LOCATIONS:
Locations (1):
- King abulaziz University, Dental University Hospital, Jeddah, P.O Box 80209, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Baik A, Alamoudi N, Felemban O, El-Housseiny A, Almabadi E, Baik K, Altuwirqi A, Masoud I. Prevention of occlusal caries using VanishTM XT: an 18-month follow-up randomized clinical trial. BMC Oral Health. 2024 Nov 1;24(1):1328. doi: 10.1186/s12903-024-05095-8. PMID 39487418